CLINICAL TRIAL: NCT07207577
Title: Evaluation of Physiological and Psychological Factors Involved in Exercise Intolerance in Patients With Transfusion-dependent β-thalassemia
Brief Title: Evaluation of Physiological and Psychological Factors Involved in Exercise Intolerance in Patients With β-TTD
Acronym: THALEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Collaborators: Université Savoie Mont Blanc (Other); Laboratoire de Psychologie et NeuroCognition (LPNC), Université Grenoble Alpes (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CHMS25002; 2025-A00051-48 (Other: ANSM)
Record Dates: First submitted 2025-09-16; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Beta Thalassemia Transfusion Dependent
Keywords: physical ability; Beta thalassemia transfusion dependent; control subjects

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): control participant without Beta thalassemia
  Interventions: Other: Maximal incremental exercise test
- Beta thalassemia transfusion dependent (Experimental): same intervention than control group
  Interventions: Other: Maximal incremental exercise test

INTERVENTIONS:
Other: Maximal incremental exercise test — Participants will perform a symptom-limited maximal incremental exercise test on a cycle ergometer.

SUMMARY:
The goal of this clinical trial is to compare physical ability of patients with transfusion-dependent β-thalassemia to control subjects. The main question it aims to answer is:

is there a difference in power output at first lactate threshold between patients with transfusion-dependent β-thalassemia and control subjects during maximal incremental exercise test.

Participants will have to realise differents exams including measurement of body compposition, maximal incremental exercise test, vertical jump, vasoreactivity test, blood sampling, quality of life questionnaires and neuromuscular assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older

  * Patients with transfusion-dependent β-thalassaemia (B0 or B+)
  * Patients who have undergone blood transfusions at intervals of between 1 and 8 weeks for at least 5 years.
  * Have given their free and informed written consent after being informed of the purpose of the study, its conduct and its risks.
  * Be affiliated with a social security scheme.
  * Not participating in any other interventional studies during the duration of this study

Control subjects must meet all of the following criteria to participate in the study:

* Subject aged 18 years or older
* Matched in age and gender to a βTTD patient included in the study.
* Declaring to be free of known acute or chronic pathologies.
* Have given their free written consent after being informed of the purpose of the study, its conduct and its risks.
* Be affiliated with a social security scheme.
* Not participate in any other interventional study during the duration of this study.
* Have 'low' or 'moderate' IPAQ results (inactive or slightly active).

Exclusion Criteria:

* - Having received a bone marrow transplant.
* History of thromboembolic disease.
* Hospitalised for cardiac decompensation in the last 12 months.
* Lack of use of limbs (amputee, paraplegic, quadriplegic)
* Unable to comply with protocol requirements for social, family or other reasons, as determined by the investigator.
* Known concomitant medical condition that could affect compliance with the protocol
* benefiting of enhanced protection, namely minors, persons deprived of their liberty by judicial or administrative decision, adults under legal protection and, finally, patients in emergency situations.
* Unable to give consent.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Power at the first lactate threshold (PSL1) collected during the maximal incremental exercise test, compared between the two groups | 7 days after a transfusion for patient
  Participants perform a maximal incremental exercise test on a cycle ergometer. The protocol includes one-minute intervals, with increments and initial power varying according to the subject's age and gender. The exercise continues until the subject is unable to maintain the power imposed by the current level. A drop of blood sample is taken from the earlobe and immediately analyzed to measure blood lactate concentration and determine first lactate threshold.

SECONDARY OUTCOMES:
Comparison of power values at lactate threshold 2 between βTTD patients and control subjects. | 7 days after a transfusion for patients
  During the exercise test, a drop of blood is taken from the earlobe and immediately analyzed to measure blood lactate concentration and determine secondlactate threshold (LT2).
Comparison between βTTD patients and control subjects of oxygen consumption efficiency slope values (OUES for Oxygen Uptake Efficiency Slope) | 7 days after a transfusion for patients
  Cardio-pulmonary parameters are measured continuously throughout the maximum incremental exercise test and are used to calculate, among other things, the oxygen uptake efficiency slope (OUES), an indicator of the subject's ability to transport and use oxygen.
Comparison between βTTD patients and control subjects of cardiac output values combining heart rate and systolic ejection volume values during maximal exercise. | 7 days after a transfusion for patients
  Values will be recorder during maximal incremental exercise test. Heart rate and systolic ejection volume values is continuously recorded by bioimpedance measurement.
Comparison of muscle mass values between βTTD patients and control subjects | 7 days after a transfusion for patients
  A body composition measurement will be performed using bioimpedance analysis.
Comparison between βTTD patients and control subjects of first-second expiratory flow values (FEV1, L) | 7 days after a transfusion for patients
  A spirometry test will be performed. After taking a deep breath, the participant will be asked to exhale as quickly as possible into the spirometer.
Comparison between βTTD patients and control subjects of maximum grip strength, jump height and reactive strength index values | 7 days after a transfusion for patients
  Jump height will be evaluate using video analysis.
Compare neuromuscular function between βTTD patients and control subjects | 7 days after a transfusion for patients
  Nerve conduction will be assessed by electroneuromyography (ENMG). Muscle electrical activity will be measured by ENMG following low-intensity electrical stimulation to collect the F wave. This test will measure: nerve conduction velocity, latency between nerve stimulation and response, response amplitude, and response duration.
Compare the level of physical activity between βTTD patients and control subjects | During inclusion visit, at day 1
  Level of activvity will be assessed with of International Physical Activity Questionnaire
Compare anxiety levels between βTTD patients and control subjects. | During second visit, occuring during a transfusion visit and no longer than 3 months after the inclusion.
  score to HADS questionnaire
Comparison between βTTD patients and control subjects of muscle reoxygenation slope values upon removal of arterial occlusion | 7 days after a transfusion for patients
  A vasoreactivity test will then be performed at rest following venous occlusion, in order to measure the ability to reoxygenate the tissue.
Correlation within the βTTD group between physical ability and cardiac iron load, hepatic iron load and EPO | 7 days after a transfusion for patients
  Correlation within the βTTD group between power at lactate threshold 1 (see primary outcome) and cardiac T2* , hepatic iron concentration and EPO level wich will be taken in patient medical file
Correlation within the βTTD group between testosterone (men) or oestrogen (women) levels and muscle mass in kg | 7 days after a transfusion for patients
  data collected in patient medical file
Correlation within the βTTD group between quality of life and physical ability | During second visit, occuring during a transfusion visit and no longer than 3 months after the inclusion.
  SF36 questionnaire will be done and scoore will be correlated to power at first lactic threshold
Assessing the link between perceived fatigue and physical activity levels in βTTD patients | During second visit, occuring during a transfusion visit and no longer than 3 months after the inclusion.
  Correlation between the score at FACIT-F questionnaires compared to scores at IPAQ questionnaires
Assessing the link between physical fitness and fatigue/pain experienced by βTTD patients | During second visit, occuring during a transfusion visit and no longer than 3 months after the inclusion.
  Correlation within the βTTD group between power at lactate threshold 1 and FACIT-F and BPI scores (multivariate analysis).
Assessing the link between microvascular vasoreactivity, inflammation and haemolysis in βTTD patients | 7 days after transfusion for patients
  Correlation within the βTTD group between the reoxygenation slope and blood concentrations of CRP, LDH, and indirect bilirubin
Assessing motivation for physical activity in βTTD patients | During second visit, occuring during a transfusion visit and no longer than 3 months after the inclusion.
  Description of the EMAPS score
Comparison between βTTD patients and control subjects of vital capacity (VC, L) | 7 days after a transfusion for patients
  A spirometry test will be performed. After taking a deep breath, the participant will be asked to exhale as quickly as possible into the spirometer.
Comparison between βTTD patients and control subjects of maximum exercise ventilation (VE, L.min-1) | 7 days after a transfusion for patients
  The ventilation rate will be continuously monitored during CPET. The ventilation rate value corresponding to the time of maximal exercise based on oxygen consumption will be used.
Comparison between βTTD patients and control subjects of maximum grip strength (kg) | 7 days after a transfusion for patients
  Maximum grip strength will be assessed with a hand dynamometer.
Comparison between βTTD patients and control subjects of reactive strength index values | 7 days after a transfusion for patients
  Reactive strength index values will be calculated based on jump height divided by the time to take-off

CONTACTS AND LOCATIONS:
Overall Officials: Laurent MESSONNIER, Study Chair — Université Savoie Mont Blanc; Pierre FAURIE, Principal Investigator — CH Metropole Savoie; Mathilde NOGUER, Study Chair — Université Savoie Mont Blanc
Locations (1):
- CH Métropole Savoie, Chambéry, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verhamme DT, Arents JC, Postma PW, Crielaard W, Hellingwerf KJ. Glucose-6-phosphate-dependent phosphoryl flow through the Uhp two-component regulatory system. Microbiology (Reading). 2001 Dec;147(Pt 12):3345-52. doi: 10.1099/00221287-147-12-3345. PMID 11739766